Tittle:

Effects of ecoguided percutaneous peroneal nerve percutaneous neuromodulation (EPNM) and neuromuscular exercise in the management of chronic ankle instability (CAI): a randomised clinical trial (RCT).

**DATE:** 19/05/2023

## **Annex 3: INFORMED CONSENT**

**STUDY TITLE:** Effects of echo-guided percutaneous neuromodulation (EPNM) of the common peroneal nerve and neuromuscular exercise in the management of chronic ankle instability (CTI).

MAIN INVESTIGATOR: Alberto Nava Varas

| CENTER: Gimbernat Cantabria University School |
|---|
| Mr./Ms <u>.</u> |
| (Name and surname of the patient in CAPITAL LETTERS) |
| I have read and understood the information sheet that has been given to me about the |
| study indicated above. I have received enough information about the study. He asked all |
| the questions he needed about the study. I have spoken with the PhD |
| studentwith whom I have clarified possible doubts. |
| I understand that my participation is voluntary. |
| I understand that I can withdraw from the study: |
| Whenever you want |
| Without giving explanations |
| Without affecting my medical care |
| I understand that the personal information I provide will remain confidential and will not |
| be disclosed to anyone without my consent. |
| I understand that my participation in the study implies authorizing |
| and I freely give my consent to participate in the study. |

## WITHDRAWAL OF CONSENT:

| Mr./Ms. | I withdraw |
|---|---|
| the consent granted for my participation in the above-mentioned study. | |
| Date and signature: | |